CLINICAL TRIAL: NCT03204786
Title: Intranasal Vasopressin Treatment in Children With Autism
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Antonio Hardan, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-39972; 1R01HD091972 (NIH)
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Results first posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-08

CONDITIONS: Autism; Autism Spectrum Disorder; ASD
Keywords: Autism Spectrum Disorder (ASD); Autism
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder | interventions — Vasopressins; Arginine Vasopressin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Vasopressin-Vasopressin (Experimental): 8 weeks of vasopressin nasal spray (16 international units twice daily)
  Interventions: Drug: Vasopressin (USP) Injectable Solution [Vasostrict]
- Placebo-Vasopressin (Experimental): 4 weeks of placebo nasal spray followed by 4 weeks of vasopressin nasal spray (16 international units twice daily)
  Interventions: Drug: Vasopressin (USP) Injectable Solution [Vasostrict]; Drug: Placebo
- Placebo-Placebo (Placebo Comparator): 8 weeks of placebo nasal spray; followed by a 4 week open-label extension of vasopressin nasal spray (16 international units twice daily)
  Interventions: Drug: Vasopressin (USP) Injectable Solution [Vasostrict]; Drug: Placebo

INTERVENTIONS:
Drug: Vasopressin (USP) Injectable Solution [Vasostrict] — Nasal Spray
Drug: Placebo — Placebo Nasal Spray
  Arms: Placebo-Placebo; Placebo-Vasopressin

SUMMARY:
The purpose of this clinical trial is to investigate the effectiveness of vasopressin nasal spray for treating symptoms associated with autism. Vasopressin is a hormone that is produced naturally within the body and has been implicated in regulating social behaviors. It has been proposed that administration of the hormone may also help improve social functioning in individuals with autism.

ELIGIBILITY:
Inclusion Criteria:

* Medically healthy outpatients between 6 and 17 years of age;
* Diagnostic and Statistical Manual 5th edition (DSM-5) criteria for Autism Spectrum Disorder (ASD) on the basis of clinical evaluation, confirmed with the Autism Diagnostic Interview Revised (ADI-R) and Autism Diagnostic Observation Schedule, Second Edition (ADOS-2) or Childhood Autism Rating Scale, Second Edition (CARS-2);
* males and females;
* intelligence quotient (IQ) of 40 and above;
* rating of 4 or higher on the Social Communication domain of the Clinical Global Impressions Severity (CGI-S);
* Social Responsiveness Scale-2 Total Score of 70 and above;
* care provider who can reliably bring participant to clinic visits, provide trustworthy ratings, and interacts with participant on a regular basis;
* stable concomitant psychotropic medications or medications potentially affecting vasopressin for at least 4 weeks (with the exception of fluoxetine, 6 weeks);
* no planned changes in psychosocial and biomedical interventions during the trial;
* willingness to provide blood samples and ability to participate in key study procedures (i.e., diagnostic assessments and laboratory safety measurements).

Exclusion Criteria:

* DSM-5 diagnosis of schizophrenia, schizoaffective disorder, or psychotic disorder;
* regular nasal obstruction or nosebleeds;
* unstable medical conditions such as migraine, asthma attacks, or seizures, and significant physical illness (e.g. serious liver disease, renal dysfunction, or cardiac pathology);
* clinically significant abnormal electrocardiogram reading;
* history of hypersensitivity to vasopressin, its analogs, or compounding preservatives (e.g., chlorobutanol);
* evidence of a genetic mutation known to cause ASD or intellectual disability (e.g., Fragile X Syndrome); or metabolic, or infectious etiology for ASD on the basis of medical history, neurologic history, and available tests for inborn errors of metabolism and chromosomal analysis;
* significant hearing or vision impairments;
* habitually drinks large volumes of water;
* pregnant or sexually active females not using a reliable method of contraception;
* current use of any medications known to interact with vasopressin including: 1) carbamazepine (i.e., Tegretol); chlorpropamide; clofibrate; urea; fludrocortisone; tricyclic antidepressants (all of which may potentiate the antidiuretic effect of vasopressin when used concurrently); 2) demeclocycline; norepinephrine; lithium; heparin; alcohol (all of which may decrease the antidiuretic effect of vasopressin when used concurrently); 3) ganglionic blocking agents including benzohexonium, chlorisondamine, pentamine (all of which may produce a marked increase in sensitivity to the pressor effects of vasopressin);
* previous participation in a vasopressin clinical trial or current use of vasopressin;
* current use of desmopressin (DDAVP) or oxytocin.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 157 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Y. Hardan, M.D., Principal Investigator — Stanford University; Karen J. Parker, Ph.D., Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
National Database for Autism Research (NDAR) Submission per NIH requirements

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized to one of three groups for two 4-week treatment periods. Participants in the Placebo-Placebo group were given the opportunity to enroll in a 4-week open-label extension period.
Pre-assignment Details: 323 participants were screened. 157 participants signed informed consent, and 108 were randomized.
Groups:
- Placebo-Placebo: 8 weeks of placebo nasal spray; followed by a 4 week optional open-label extension of vasopressin nasal spray (16 international units twice daily)
Period: Treatment Period 1 (4 Weeks)
Arm/Group | Vasopressin-Vasopressin | Placebo-Vasopressin | Placebo-Placebo
Started | 23 | 46 | 39
Received Intervention | 23 | 44 | 39
Completed | 22 | 41 | 39
Not Completed | 1 | 5 | 0
Period: Treatment Period 2 (4 Weeks)
Arm/Group | Vasopressin-Vasopressin | Placebo-Vasopressin | Placebo-Placebo
Started | 21 | 38 | 39
Completed | 19 | 38 | 36
Not Completed | 2 | 0 | 3
Period: Open-label Extension (4 Weeks)
Arm/Group | Vasopressin-Vasopressin | Placebo-Vasopressin | Placebo-Placebo
Started | 0 | 0 | 32
Completed | 0 | 0 | 29
Not Completed | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: Participants who were randomized and treated (received intervention)
Groups:
- Total: Total of all reporting groups
Arm/Group | Vasopressin-Vasopressin | Placebo-Vasopressin | Placebo-Placebo | Total
Number analyzed (Participants) | 23 | 44 | 39 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.35 (3.24) | 10.41 (3.23) | 10.72 (3.5) | 10.51 (3.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 5 | 14
  Male | 20 | 38 | 34 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 8 | 9 | 21
  Not Hispanic or Latino | 17 | 31 | 27 | 75
  Unknown or Not Reported | 2 | 5 | 3 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4 | 11 | 15 | 30
  Black | 0 | 2 | 1 | 3
  Multiracial | 3 | 6 | 3 | 12
  Other | 2 | 5 | 4 | 11
  Unknown | 2 | 1 | 0 | 3
  White | 12 | 19 | 16 | 47
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 44 | 39 | 106

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Parent Rated Social Responsiveness Scale, Second Edition (SRS-2) Total Scores During Treatment.
Description: Social Responsiveness Scale, 2nd Edition (SRS) scores measure social abilities with lower scores meaning better social abilities. The SRS-2 is reported as a total score (T-Score Range: 37 to above 90), and the Diagnostic and Statistical Manual of Mental Disorders (DSM)-5-compatible Social Communication and Interaction (SCI) score (T-Score Range: 36 to above 90) and Restricted Interests and Repetitive Behavior (RRB) score (T-Score range: 41 to above 90). A T-score of 50 indicates the population mean with a standard deviation of 10. Higher scores correspond to greater symptom levels (≤ 59: within normal limits; 60-65: mild range; 66-75: moderate range; ≥ 76: severe range). Change is reported as 4-week minus the baseline score, and 8-week minus the 4-week score. For this outcome, the baseline score is the average of the screening visit and baseline visit (average approximately 2 to 3 weeks after the screening visit).
Time Frame: baseline, 4-week, 8-week
Population: Participants with available data at the respective time point
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Vasopressin-Vasopressin | Placebo-Vasopressin | Placebo-Placebo
Number analyzed (Participants) | 22 | 41 | 39
T-score
  Total score - baseline | 81.3690 (2.1052) | 79.6795 (1.5448) | 82.2281 (1.5650)
  Total score - change from baseline at 4-week | -5.6779 (1.6830) | -4.5448 (1.2298) | -6.4832 (1.2695)
  Total score - 4-week | 75.0000 (2.1052) | 74.7821 (1.5448) | 74.8816 (1.5650)
  Total score - change from week 4 at week 8: number analyzed (Participants) | 19 | 38 | 36
  Total score - change from week 4 at week 8 | -3.4420 (1.7758) | -5.3854 (1.2964) | -1.0443 (1.3267)
  SCI score - baseline | 81.2500 (2.0892) | 79.3333 (1.5330) | 81.5987 (1.5531)
  SCI score - change from baseline at 4-week | -5.6451 (1.6475) | -4.6366 (1.2024) | -6.3462 (1.2385)
  SCI score - 4-week | 74.9405 (2.0892) | 74.3718 (1.5330) | 74.5263 (1.5531)
  SCI score - change from week 4 at week 8: number analyzed (Participants) | 19 | 38 | 36
  SCI score - change from week 4 at week 8 | -2.8205 (1.7326) | -5.1550 (1.2689) | -0.9782 (1.2962)
  RRB score - baseline | 78.0000 (2.3077) | 77.0128 (1.6934) | 80.4408 (1.7155)
  RRB score - change from baseline at 4-week | -5.4830 (1.8580) | -3.5584 (1.3617) | -6.2517 (1.4083)
  RRB score - 4-week | 71.8095 (2.3077) | 73.0641 (1.6934) | 72.6974 (1.7155)
  RRB score - change from week 4 at week 8: number analyzed (Participants) | 19 | 38 | 36
  RRB score - change from week 4 at week 8 | -5.4995 (1.9770) | -5.4625 (1.4287) | -0.9253 (1.4705)

2. Secondary Outcome: Change From Baseline in Clinical Global Impression (CGI) Scores During Treatment.
Description: Clinician assessment of CGI severity (CGI-S) and CGI improvement (CGI-I) scores.
  * Higher scores on the CGI-S mean greater social and communication deficits (range: 1 to 7).
  * Lower scores on the CGI-I correspond to greater improvement in the areas assessed in the CGI-S, and higher scores correspond to worsening (range: 1 to 7). There is no baseline score for the CGI-I, it represents the clinician's subjective assessment of change.
Time Frame: baseline; 4-week; 8-week
Population: Participants with data at the respective time point
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Vasopressin-Vasopressin | Placebo-Vasopressin | Placebo-Placebo
Number analyzed (Participants) | 22 | 41 | 39
score on a scale
  CGI-S score - baseline | 4.8182 (0.1206) | 4.6585 (0.08834) | 4.7692 (0.09058)
  CGI-S score - change from baseline at 4-week | 0.001903 (0.03413) | -0.00113 (0.02499) | -0.02467 (0.02562)
  CGI-S score - 4-week | 4.8177 (0.1209) | 4.6576 (0.08846) | 4.7416 (0.09070)
  CGI-S score - change from 4-week at 8-week: number analyzed (Participants) | 19 | 38 | 36
  CGI-S score - change from 4-week at 8-week | -0.05149 (0.03633) | -0.00254 (0.02589) | -0.02795 (0.02651)
  CGI-I: 4-week (end of treatment period 1) | 3.8636 (0.1132) | 3.7073 (0.08293) | 3.8205 (0.08503)
  CGI-I: 8-week (end of treatment period 2): number analyzed (Participants) | 19 | 38 | 36
  CGI-I: 8-week (end of treatment period 2) | 3.5892 (0.1200) | 3.5899 (0.08547) | 3.7307 (0.08777)

3. Secondary Outcome: Change From Baseline on Reading the Mind in the Eyes Test (RMET) During Treatment.
Description: Score range: 0 to 28; higher scores mean better ability to read emotions and lower scores mean worse ability to read emotions.
Time Frame: baseline; 4-week; 8-week
Population: Participants with data at the respective time point
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Vasopressin-Vasopressin | Placebo-Vasopressin | Placebo-Placebo
Number analyzed (Participants) | 23 | 46 | 39
score on a scale
  Baseline: number analyzed (Participants) | 9 | 20 | 19
  Baseline | 16.5556 (1.8377) | 14.7222 (1.2995) | 15.5789 (1.2648)
  Change from baseline at 4-week: number analyzed (Participants) | 9 | 18 | 19
  Change from baseline at 4-week | 1.6440 (1.2030) | -0.02870 (0.8518) | -0.4319 (0.8267)
  4-week: number analyzed (Participants) | 9 | 18 | 19
  4-week | 18.3273 (1.9019) | 14.8889 (1.2995) | 15.2876 (1.3064)
  Change from 4-week at 8-week: number analyzed (Participants) | 8 | 18 | 17
  Change from 4-week at 8-week | -0.2844 (1.3008) | 0.5628 (0.8510) | -0.2156 (0.8771)

4. Secondary Outcome: Change From Baseline on the Facial Emotion Recognition Test During Treatment.
Description: Score range: 0 to 42; higher scores mean better facial emotion recognition abilities. Lower scores mean worse facial emotion recognition abilities.
Time Frame: baseline; 4-week; 8-week
Population: Participants with data at the respective time point
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Vasopressin-Vasopressin | Placebo-Vasopressin | Placebo-Placebo
Number analyzed (Participants) | 23 | 46 | 39
score on a scale
  Baseline | 25.2667 (1.9330) | 30.3913 (1.5610) | 31.3333 (1.6336)
  Change from baseline at 4-week: number analyzed (Participants) | 15 | 23 | 21
  Change from baseline at 4-week | 0.05134 (1.0362) | 0.2458 (0.8136) | -0.1705 (0.8543)
  4-week: number analyzed (Participants) | 15 | 23 | 21
  4-week | 26.3341 (1.9736) | 30.3846 (1.5814) | 30.7990 (1.6449)
  Change from 4-week at 8-week: number analyzed (Participants) | 13 | 21 | 20
  Change from 4-week at 8-week | 2.3733 (1.0904) | -0.5105 (0.8605) | 1.7945 (0.8736)

5. Secondary Outcome: Change From Baseline in Parent Rated Repetitive Behavior Scale Revised (RBS-R) Scores During Treatment.
Description: Score range: 0 to 129; higher scores on the RBS-R mean higher levels of repetitive and restricted behaviors.
Time Frame: baseline; 4-week; 8-week
Population: Participants with data at the respective time point
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Vasopressin-Vasopressin | Placebo-Vasopressin | Placebo-Placebo
Number analyzed (Participants) | 23 | 46 | 39
score on a scale
  Baseline | 24.9872 (3.8628) | 26.4763 (2.9263) | 32.6154 (2.8720)
  Change from baseline at 4-week: number analyzed (Participants) | 21 | 37 | 39
  Change from baseline at 4-week | -1.4292 (2.4939) | -4.6282 (1.8785) | -5.4530 (1.8509)
  4-week: number analyzed (Participants) | 21 | 37 | 39
  4-week | 22.7130 (4.0020) | 21.4958 (2.9623) | 27.9896 (2.9411)
  Change from 4-week at 8-week: number analyzed (Participants) | 18 | 35 | 35
  Change from 4-week at 8-week | -4.5054 (2.6993) | -2.1610 (1.9440) | -0.08268 (1.9332)

6. Secondary Outcome: Change From Baseline in Parent Rated Spence Children's Anxiety Scale (SCAS) During Treatment.
Description: Scale measuring severity of anxiety symptoms. Score range: 0 to 114; higher scores mean higher levels of anxiety, lower scores mean lower levels of anxiety.
Time Frame: baseline; 4-week; 8-week
Population: Participants with data at the respective time point
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Vasopressin-Vasopressin | Placebo-Vasopressin | Placebo-Placebo
Number analyzed (Participants) | 23 | 46 | 39
score on a scale
  Baseline | 18.9944 (2.3258) | 16.0513 (1.6862) | 17.4681 (1.6970)
  Change from baseline at 4-week: number analyzed (Participants) | 20 | 39 | 35
  Change from baseline at 4-week | -2.1798 (1.4413) | -2.5005 (1.0257) | -2.5485 (1.0439)
  4-week: number analyzed (Participants) | 20 | 39 | 38
  4-week | 14.7648 (2.3563) | 14.0044 (1.7201) | 13.8016 (1.7202)
  Change from 4-week at 8-week: number analyzed (Participants) | 19 | 36 | 36
  Change from 4-week at 8-week | -3.1160 (1.4720) | -3.9195 (1.0731) | -1.1805 (1.0743)

7. Secondary Outcome: Change From Baseline on Electrocardiogram (EKG) P Duration During Treatment.
Time Frame: baseline to 4-week, 8-week, and 12-week
Population: Participants with available data at the respective time point
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Vasopressin-Vasopressin | Placebo-Vasopressin | Placebo-Placebo
Number analyzed (Participants) | 23 | 46 | 39
milliseconds
  Baseline | 87.9 (1.88) | 86.5 (1.53) | 86.7 (1.18)
  4-weeks (end of treatment period 1): number analyzed (Participants) | 22 | 41 | 39
  4-weeks (end of treatment period 1) | 83.7 (2.11) | 87.1 (1.88) | 87.0 (1.44)
  8-weeks (end of treatment period 2): number analyzed (Participants) | 19 | 38 | 36
  8-weeks (end of treatment period 2) | 88.2 (2.03) | 85.6 (1.5) | 84.4 (1.36)
  12-weeks (end of open-label extension): number analyzed (Participants) | 0 | 0 | 29
  12-weeks (end of open-label extension) |  |  | 89.6 (1.33)

8. Secondary Outcome: Change From Baseline on Electrocardiogram (EKG) PR Interval During Treatment.
Time Frame: baseline to 4-week, 8-week, and 12-week
Population: Participants with available data at the respective time point
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Vasopressin-Vasopressin | Placebo-Vasopressin | Placebo-Placebo
Number analyzed (Participants) | 23 | 46 | 39
milliseconds
  Baseline | 136 (3.48) | 138 (2.38) | 137 (2.34)
  4-weeks (end of treatment period 1): number analyzed (Participants) | 22 | 41 | 39
  4-weeks (end of treatment period 1) | 136 (3.48) | 139 (3.02) | 140 (2.6)
  8-weeks (end of treatment period 2): number analyzed (Participants) | 19 | 38 | 36
  8-weeks (end of treatment period 2) | 135 (2.96) | 141 (.345) | 139 (2.95)
  12-weeks (end of open-label extension): number analyzed (Participants) | 0 | 0 | 29
  12-weeks (end of open-label extension) |  |  | 142 (2.73)

9. Secondary Outcome: Change From Baseline on Electrocardiogram (EKG) QRS Interval During Treatment.
Time Frame: baseline to 4-week, 8-week, and 12-week
Population: Participants with available data at the respective time point
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Vasopressin-Vasopressin | Placebo-Vasopressin | Placebo-Placebo
Number analyzed (Participants) | 23 | 46 | 39
milliseconds
  Baseline | 87.3 (1.76) | 89.5 (1.27) | 86.7 (1.44)
  4-weeks (end of treatment period 1): number analyzed (Participants) | 22 | 41 | 39
  4-weeks (end of treatment period 1) | 89.5 (2.45) | 88.6 (41.5) | 86.5 (1.24)
  8-weeks (end of treatment period 2): number analyzed (Participants) | 19 | 38 | 36
  8-weeks (end of treatment period 2) | 29.3 (0.87) | 89.2 (1.52) | 86.2 (1.7)
  12-weeks (end of open-label extension): number analyzed (Participants) | 0 | 0 | 29
  12-weeks (end of open-label extension) |  |  | 84.6 (1.52)

10. Secondary Outcome: Change From Baseline on Electrocardiogram (EKG) QT Interval During Treatment.
Time Frame: baseline to 4-week, 8-week, and 12-week
Population: Participants with available data at the respective time point
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Vasopressin-Vasopressin | Placebo-Vasopressin | Placebo-Placebo
Number analyzed (Participants) | 23 | 46 | 39
milliseconds
  Baseline | 399 (6.03) | 355 (3.61) | 348 (4.05)
  4-weeks (end of treatment period 1): number analyzed (Participants) | 22 | 41 | 39
  4-weeks (end of treatment period 1) | 352 (6.94) | 365 (4.24) | 350 (4.27)
  8-weeks (end of treatment period 2): number analyzed (Participants) | 19 | 38 | 36
  8-weeks (end of treatment period 2) | 355 (5.37) | 359 (4.79) | 354 (5.23)
  12-weeks (end of open-label extension): number analyzed (Participants) | 0 | 0 | 29
  12-weeks (end of open-label extension) |  |  | 344 (4.00)

11. Secondary Outcome: Change From Baseline on Blood Clinical Labs (Sodium) During Treatment.
Time Frame: baseline to 4-week, 8-week, and 12-week
Population: Participants with available data at the respective time point
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Vasopressin-Vasopressin | Placebo-Vasopressin | Placebo-Placebo
Number analyzed (Participants) | 23 | 46 | 39
mmol/L
  Baseline | 139 (0.457) | 139 (0.252) | 139 (0.434)
  4-weeks (end of treatment period 1): number analyzed (Participants) | 22 | 41 | 39
  4-weeks (end of treatment period 1) | 139 (0.434) | 139 (0.293) | 139 (0.232)
  8-weeks (end of treatment period 2): number analyzed (Participants) | 19 | 38 | 36
  8-weeks (end of treatment period 2) | 140 (0.402) | 139 (0.426) | 139 (0.34)
  12-weeks (end of open-label extension): number analyzed (Participants) | 0 | 0 | 29
  12-weeks (end of open-label extension) |  |  | 139 (0.291)

12. Secondary Outcome: Change From Baseline on Blood Clinical Labs (Potassium) During Treatment.
Time Frame: baseline to 4-week, 8-week, and 12-week
Population: Participants with available data at the respective time point
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Vasopressin-Vasopressin | Placebo-Vasopressin | Placebo-Placebo
Number analyzed (Participants) | 23 | 46 | 39
mmol/L
  Baseline | 4.07 (0.0661) | 4.14 (0.0497) | 4.21 (0.0564)
  4-weeks (end of treatment period 1): number analyzed (Participants) | 22 | 41 | 39
  4-weeks (end of treatment period 1) | 4.07 (0.0374) | 4.13 (0.049) | 4.3 (0.0751)
  8-weeks (end of treatment period 2): number analyzed (Participants) | 19 | 38 | 36
  8-weeks (end of treatment period 2) | 4.16 (0.0922) | 4.17 (0.0714) | 4.24 (0.0859)
  12-weeks (end of open-label extension): number analyzed (Participants) | 0 | 0 | 29
  12-weeks (end of open-label extension) |  |  | 4.12 (0.0742)

13. Secondary Outcome: Change From Baseline on Blood Clinical Labs (Chloride) During Treatment.
Description: Change from baseline on blood clinical labs (Chloride) during treatment.
Time Frame: baseline to 4-week, 8-week, and 12-week
Population: Participants with available data at the respective time point
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Vasopressin-Vasopressin | Placebo-Vasopressin | Placebo-Placebo
Number analyzed (Participants) | 23 | 46 | 39
mmol/L
  Baseline | 103 (0.375) | 103 (0.298) | 102 (0.291)
  4-weeks (end of treatment period 1): number analyzed (Participants) | 22 | 41 | 39
  4-weeks (end of treatment period 1) | 103 (0.502) | 103 (0.305) | 103 (0.296)
  8-weeks (end of treatment period 2): number analyzed (Participants) | 19 | 38 | 36
  8-weeks (end of treatment period 2) | 103 (0.501) | 102 (0.362) | 102 (0.313)
  12-weeks (end of open-label extension): number analyzed (Participants) | 0 | 0 | 29
  12-weeks (end of open-label extension) |  |  | 102 (0.308)

14. Secondary Outcome: Change From Baseline on Blood Clinical Labs (CO2) During Treatment.
Time Frame: baseline to 4-week, 8-week, and 12-week
Population: Participants with available data at the respective time point
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Vasopressin-Vasopressin | Placebo-Vasopressin | Placebo-Placebo
Number analyzed (Participants) | 23 | 46 | 39
mmol/L
  Baseline | 25 (0.574) | 25.1 (0.273) | 25.2 (0.279)
  4-weeks (end of treatment period 1): number analyzed (Participants) | 22 | 41 | 39
  4-weeks (end of treatment period 1) | 25.5 (0.515) | 25.3 (0.291) | 25.7 (0.452)
  8-weeks (end of treatment period 2): number analyzed (Participants) | 19 | 38 | 36
  8-weeks (end of treatment period 2) | 25.8 (0.505) | 24.8 (0.321) | 25.3 (0.374)
  12-weeks (end of open-label extension): number analyzed (Participants) | 0 | 0 | 29
  12-weeks (end of open-label extension) |  |  | 25 (0.362)

15. Secondary Outcome: Change From Baseline on Blood Clinical Labs (Anion Gap) During Treatment.
Time Frame: baseline to 4-week, 8-week, and 12-week
Population: Participants with available data at the respective time point
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Vasopressin-Vasopressin | Placebo-Vasopressin | Placebo-Placebo
Number analyzed (Participants) | 23 | 46 | 39
mmol/L
  Baseline | 11.3 (0.524) | 11.6 (0.291) | 11 (0.34)
  4-weeks (end of treatment period 1): number analyzed (Participants) | 22 | 41 | 39
  4-weeks (end of treatment period 1) | 11 (0.439) | 11.1 (0.384) | 10.8 (0.482)
  8-weeks (end of treatment period 2): number analyzed (Participants) | 19 | 38 | 36
  8-weeks (end of treatment period 2) | 10.8 (0.763) | 11.6 (0.34) | 11.5 (0.479)
  12-weeks (end of open-label extension): number analyzed (Participants) | 0 | 0 | 29
  12-weeks (end of open-label extension) |  |  | 10.9 (0.446)

16. Secondary Outcome: Change From Baseline on Blood Clinical Labs (Glucose) During Treatment.
Time Frame: baseline to 4-week, 8-week, and 12-week
Population: Participants with available data at the respective time point
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Vasopressin-Vasopressin | Placebo-Vasopressin | Placebo-Placebo
Number analyzed (Participants) | 23 | 46 | 39
mg/dL
  Baseline | 95.7 (2.75) | 94.4 (1.85) | 94.9 (2.21)
  4-weeks (end of treatment period 1): number analyzed (Participants) | 22 | 41 | 39
  4-weeks (end of treatment period 1) | 99 (2.8) | 93.7 (2.33) | 94.8 (2.29)
  8-weeks (end of treatment period 2): number analyzed (Participants) | 19 | 38 | 36
  8-weeks (end of treatment period 2) | 93.5 (1.31) | 94.2 (2.25) | 94.5 (2.27)
  12-weeks (end of open-label extension): number analyzed (Participants) | 0 | 0 | 29
  12-weeks (end of open-label extension) |  |  | 97 (2.84)

17. Secondary Outcome: Change From Baseline on Blood Clinical Labs (Creatinine) During Treatment.
Time Frame: baseline to 4-week, 8-week, and 12-week
Population: Participants with available data at the respective time point
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Vasopressin-Vasopressin | Placebo-Vasopressin | Placebo-Placebo
Number analyzed (Participants) | 23 | 46 | 39
mg/dL
  Baseline | 0.473 (0.0297) | 0.502 (0.0243) | 0.515 (0.0257)
  4-weeks (end of treatment period 1): number analyzed (Participants) | 22 | 41 | 39
  4-weeks (end of treatment period 1) | 0.505 (0.037) | 0.503 (0.0256) | 0.523 (0.0294)
  8-weeks (end of treatment period 2): number analyzed (Participants) | 19 | 38 | 36
  8-weeks (end of treatment period 2) | 0.531 (0.048) | 0.508 (0.0273) | 0.517 (0.0258)
  12-weeks (end of open-label extension): number analyzed (Participants) | 0 | 0 | 29
  12-weeks (end of open-label extension) |  |  | 0.5 (0.0257)

18. Secondary Outcome: Change From Baseline on Blood Clinical Labs (Urea Nitrogen) During Treatment.
Time Frame: baseline to 4-week, 8-week, and 12-week
Population: Participants with available data at the respective time point
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Vasopressin-Vasopressin | Placebo-Vasopressin | Placebo-Placebo
Number analyzed (Participants) | 23 | 46 | 39
mg/dL
  Baseline | 12.8 (0.691) | 13.7 (0.462) | 13.7 (0.465)
  4-weeks (end of treatment period 1): number analyzed (Participants) | 22 | 41 | 39
  4-weeks (end of treatment period 1) | 12.6 (0.827) | 13.4 (0.588) | 13.4 (0.587)
  8-weeks (end of treatment period 2): number analyzed (Participants) | 19 | 38 | 36
  8-weeks (end of treatment period 2) | 14.2 (0.957) | 12.2 (0.618) | 14 (0.683)
  12-weeks (end of open-label extension): number analyzed (Participants) | 0 | 0 | 29
  12-weeks (end of open-label extension) |  |  | 13.8 (0.638)

19. Secondary Outcome: Change From Baseline on Blood Clinical Labs (Calcium) During Treatment.
Time Frame: baseline to 4-week, 8-week, and 12-week
Population: Participants with available data at the respective time point
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Vasopressin-Vasopressin | Placebo-Vasopressin | Placebo-Placebo
Number analyzed (Participants) | 23 | 46 | 39
mg/dL
  Baseline | 9.45 (0.0797) | 9.54 (0.0443) | 9.55 (0.0673)
  4-weeks (end of treatment period 1): number analyzed (Participants) | 22 | 41 | 39
  4-weeks (end of treatment period 1) | 9.5 (0.0809) | 9.57 (0.0564) | 9.62 (0.0492)
  8-weeks (end of treatment period 2): number analyzed (Participants) | 19 | 38 | 36
  8-weeks (end of treatment period 2) | 9.67 (0.0642) | 9.6 (0.0671) | 9.67 (0.0568)
  12-weeks (end of open-label extension): number analyzed (Participants) | 0 | 0 | 29
  12-weeks (end of open-label extension) |  |  | 9.85 (0.058)

20. Secondary Outcome: Change From Baseline on Blood Clinical Labs (Osmolality) During Treatment.
Time Frame: baseline to 4-week, 8-week, and 12-week
Population: Participants with available data at the respective time point
Measure: Mean (Standard Error); unit: mOsm/kg
Arm/Group | Vasopressin-Vasopressin | Placebo-Vasopressin | Placebo-Placebo
Number analyzed (Participants) | 23 | 46 | 39
mOsm/kg
  Baseline | 289 (1.03) | 289 (0.735) | 290 (1.03)
  4-weeks (end of treatment period 1): number analyzed (Participants) | 22 | 41 | 39
  4-weeks (end of treatment period 1) | 289 (1.19) | 289 (0.839) | 291 (1.13)
  8-weeks (end of treatment period 2): number analyzed (Participants) | 19 | 38 | 36
  8-weeks (end of treatment period 2) | 291 (1.28) | 288 (0.937) | 290 (0.935)
  12-weeks (end of open-label extension): number analyzed (Participants) | 0 | 0 | 29
  12-weeks (end of open-label extension) |  |  | 290 (1.29)

21. Secondary Outcome: Change From Baseline on Urine Clinical Labs (Osmolality) During Treatment.
Time Frame: baseline to 4-week, 8-week, and 12-week
Population: Participants with available data at the respective time point
Measure: Mean (Standard Error); unit: mOsm/kg
Arm/Group | Vasopressin-Vasopressin | Placebo-Vasopressin | Placebo-Placebo
Number analyzed (Participants) | 23 | 46 | 39
mOsm/kg
  Baseline | 757 (72.6) | 843 (38.2) | 827 (47.3)
  4-weeks (end of treatment period 1): number analyzed (Participants) | 22 | 41 | 39
  4-weeks (end of treatment period 1) | 758 (70.3) | 810 (44.8) | 815 (45.5)
  8-weeks (end of treatment period 2): number analyzed (Participants) | 19 | 38 | 36
  8-weeks (end of treatment period 2) | 834 (68.3) | 732 (48.1) | 838 (47.9)
  12-weeks (end of open-label extension): number analyzed (Participants) | 0 | 0 | 29
  12-weeks (end of open-label extension) |  |  | 875 (60.1)

22. Secondary Outcome: Change From Baseline on Vital Signs (Systolic Blood Pressure) During Treatment.
Time Frame: Up to 12 weeks
Population: Participants with available data at the respective time point
Measure: Mean (Standard Error); unit: mmHg
Groups:
- Vasopressin-Vasopressin Group - Treatment Period 1: Parameter assessed in the Vasopressin-Vasopressin group during the first 4-week treatment period (while receiving active drug).
- Placebo-Vasopressin Group - Treatment Period 1: Parameter assessed in the Placebo-Vasopressin group during the first 4-week treatment period (while receiving placebo).
- Placebo-Placebo Group - Treatment Period 1: Parameter assessed in the Placebo-Placebo group during the first 4-week treatment period (while receiving placebo).
- Vasopressin-Vasopressin Group - Treatment Period 2: Parameter assessed in the Vasopressin-Vasopressin group during the second 4-week treatment period (while receiving active drug).
- Placebo-Vasopressin Group - Treatment Period 2: Parameter assessed in the Placebo-Vasopressin group during the second 4-week treatment period (while receiving active drug).
- Placebo-Placebo Group - Treatment Period 2: Parameter assessed in the Placebo-Placebo group during the second 4-week treatment period (while receiving placebo).
- Open-label Vasopressin: Parameter assessed in the Placebo-Placebo group during the open-label extension (after the 2 initial treatment periods, while receiving active drug).
Arm/Group | Vasopressin-Vasopressin Group - Treatment Period 1 | Placebo-Vasopressin Group - Treatment Period 1 | Placebo-Placebo Group - Treatment Period 1 | Vasopressin-Vasopressin Group - Treatment Period 2 | Placebo-Vasopressin Group - Treatment Period 2 | Placebo-Placebo Group - Treatment Period 2 | Open-label Vasopressin
Number analyzed (Participants) | 22 | 41 | 39 | 19 | 38 | 36 | 29
mmHg
  Sitting | 114 (2.78) | 107 (2.38) | 112 (1.58) | 111 (3.32) | 109 (2.22) | 110 (1.96) | 111 (2.03)
  Standing | 110 (2.13) | 109 (1.99) | 111 (1.71) | 108 (2.44) | 107 (1.79) | 112 (2.47) | 113 (2.13)
  Change from standing to sitting | -3.25 (2.16) | 1.47 (1.67) | -1.00 (1.44) | -4.06 (3.86) | -2.53 (1.34) | 1.47 (1.69) | 2.04 (1.71)

23. Secondary Outcome: Change From Baseline on Vital Signs (Diastolic Blood Pressure) During Treatment.
Time Frame: Up to 12 weeks
Population: Participants with available data at the respective time point
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Vasopressin-Vasopressin Group - Treatment Period 1 | Placebo-Vasopressin Group - Treatment Period 1 | Placebo-Placebo Group - Treatment Period 1 | Vasopressin-Vasopressin Group - Treatment Period 2 | Placebo-Vasopressin Group - Treatment Period 2 | Placebo-Placebo Group - Treatment Period 2 | Open-label Vasopressin
Number analyzed (Participants) | 22 | 41 | 39 | 19 | 38 | 36 | 29
mmHg
  Sitting | 65.8 (3.47) | 63.4 (1.34) | 67.2 (1.79) | 69.3 (3.75) | 63.6 (1.42) | 66.9 (1.75) | 65.1 (2.11)
  Standing | 70.7 (3.08) | 62.3 (1.72) | 67.0 (1.57) | 68.8 (1.41) | 65.5 (1.58) | 66.6 (1.96) | 67.8 (1.80)
  Change from standing to sitting | 4.90 (3.02) | -1.11 (1.84) | 0.167 (1.60) | -1.00 (3.96) | 1.72 (1.59) | -0.118 (2.11) | 2.65 (2.49)

24. Secondary Outcome: Change From Baseline on Vital Signs (Pulse) During Treatment.
Time Frame: Up to 12 weeks
Population: Participants with available data at the respective time point
Measure: Mean (Standard Error); unit: beats per minute (BPM)
Arm/Group | Vasopressin-Vasopressin Group - Treatment Period 1 | Placebo-Vasopressin Group - Treatment Period 1 | Placebo-Placebo Group - Treatment Period 1 | Vasopressin-Vasopressin Group - Treatment Period 2 | Placebo-Vasopressin Group - Treatment Period 2 | Placebo-Placebo Group - Treatment Period 2 | Open-label Vasopressin
Number analyzed (Participants) | 22 | 41 | 39 | 19 | 38 | 36 | 29
beats per minute (BPM)
  Sitting | 88.4 (3.40) | 84.2 (2.11) | 94.3 (2.45) | 89.2 (4.06) | 90.0 (2.95) | 90.7 (2.40) | 94.9 (3.95)
  Standing | 99.6 (3.02) | 94.8 (2.39) | 103 (2.43) | 100 (4.01) | 102 (2.91) | 105 (3.44) | 107 (3.98)
  Change from standing to sitting | 11.2 (2.25) | 10.6 (1.37) | 10.1 (1.65) | 10.9 (2.29) | 11.9 (1.77) | 14.2 (2.41) | 11.2 (2.84)

25. Secondary Outcome: Change From Baseline on Height During Treatment.
Time Frame: baseline to 4-week, 8-week, and 12-week
Population: Participants with available data at the respective time point
Measure: Mean (Standard Error); unit: cm
Arm/Group | Vasopressin-Vasopressin | Placebo-Vasopressin | Placebo-Placebo
Number analyzed (Participants) | 23 | 46 | 39
cm
  Baseline | 145 (3.91) | 146 (2.98) | 145 (2.78)
  4-weeks (end of treatment period 1): number analyzed (Participants) | 22 | 41 | 39
  4-weeks (end of treatment period 1) | 142 (5.96) | 148 (3.21) | 146 (2.76)
  8-weeks (end of treatment period 2): number analyzed (Participants) | 19 | 38 | 36
  8-weeks (end of treatment period 2) | 145 (4.43) | 148 (3.22) | 146 (2.68)
  12-weeks (end of open-label extension): number analyzed (Participants) | 0 | 0 | 29
  12-weeks (end of open-label extension) |  |  | 145 (3.26)

26. Secondary Outcome: Change From Baseline on Weight During Treatment.
Time Frame: baseline to 4-week, 8-week, and 12-week
Population: Participants with available data at the respective time point
Measure: Mean (Standard Error); unit: kg
Arm/Group | Vasopressin-Vasopressin | Placebo-Vasopressin | Placebo-Placebo
Number analyzed (Participants) | 23 | 46 | 39
kg
  Baseline | 43.2 (3.92) | 45.2 (4.24) | 45.7 (3.15)
  4-weeks (end of treatment period 1): number analyzed (Participants) | 22 | 41 | 39
  4-weeks (end of treatment period 1) | 43.9 (4.47) | 46.6 (4.92) | 46.6 (3.17)
  8-weeks (end of treatment period 2): number analyzed (Participants) | 19 | 38 | 36
  8-weeks (end of treatment period 2) | 43.0 (4.83) | 44.0 (3.38) | 46.8 (3.22)
  12-weeks (end of open-label extension): number analyzed (Participants) | 0 | 0 | 29
  12-weeks (end of open-label extension) |  |  | 47.6 (4.34)

27. Secondary Outcome: Change From Baseline on the Dosage Record Treatment Emergent Symptom Scale (DOTES) During Treatment.
Description: The DOTES evaluates a subset of symptoms related to various medical conditions. The clinician assesses intensity (0=Not assessed, 1=Not present, 2=Mild, 3=Moderate, 4=Severe), relatedness (0=None, 1=Remote, 2=Possible, 3=Probable, 4=Defined), and action taken (0=None, 1=Increased , 2=Contractive Rx, 3=Change Dose, 4=Change Dose Plus Contractive Rx, 5=Suspend Rx, 6=Discontinue Rx). Side effects are included that have increased in severity, become more likely to be related, or require action. Change from baseline is reported as the number of participants with change in these side effects during treatment.
Time Frame: Up to 12 weeks
Population: Participants with available data at the respective time point
Measure: Count of Participants; unit: Participants
Arm/Group | Vasopressin-Vasopressin Group - Treatment Period 1 | Placebo-Vasopressin Group - Treatment Period 1 | Placebo-Placebo Group - Treatment Period 1 | Vasopressin-Vasopressin Group - Treatment Period 2 | Placebo-Vasopressin Group - Treatment Period 2 | Placebo-Placebo Group - Treatment Period 2 | Open-label Vasopressin
Number analyzed (Participants) | 22 | 42 | 39 | 21 | 38 | 39 | 32
Participants
  Dizziness | 0 | 1 | 1 | 0 | 0 | 0 | 1
  Constipation | 2 | 0 | 4 | 2 | 4 | 1 | 0
  Diarrhea | 0 | 2 | 3 | 1 | 2 | 1 | 0
  Dry Mouth | 0 | 2 | 0 | 0 | 1 | 0 | 0
  Saliva Hypersecretion | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Vomiting or Nausea | 0 | 1 | 1 | 0 | 2 | 3 | 1
  Decreased Appetite | 0 | 3 | 1 | 1 | 2 | 0 | 0
  Increased Appetite | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Agitation | 2 | 3 | 3 | 2 | 2 | 3 | 1
  Headache | 2 | 4 | 3 | 0 | 5 | 4 | 4
  Initial Insomnia | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Middle Insomnia | 0 | 0 | 0 | 0 | 1 | 1 | 0
  Unspecified Insomnia | 0 | 3 | 0 | 0 | 2 | 0 | 0
  Aggression | 1 | 8 | 10 | 5 | 8 | 7 | 8
  Depressed Mood | 1 | 1 | 2 | 2 | 1 | 1 | 1
  Hyperactivity | 0 | 4 | 1 | 0 | 1 | 0 | 1
  Nasal Congestion | 2 | 6 | 13 | 5 | 6 | 10 | 7
  Pruritus | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Rash | 0 | 3 | 2 | 1 | 3 | 2 | 1

28. Secondary Outcome: Change From Baseline in Overt Aggression Scale (OAS) During Treatment.
Time Frame: 2-week, 4-week; 6-week, 8-week
Reporting Status: Not Posted

29. Secondary Outcome: Baseline Vasopressin Concentration Predicting Primary and Secondary Behavioral Outcome Measures.
Time Frame: 4-week; 8-week
Reporting Status: Not Posted

30. Secondary Outcome: Adverse Event Severity
Description: Adverse events collated according to intensity for each pre-allocated treatment group.
Time Frame: Up to 12 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Vasopressin-Vasopressin Group - Treatment Period 1: Adverse events occurring in the Vasopressin-Vasopressin group during the first 4-week treatment period (while receiving active drug).
- Placebo-Vasopressin Group - Treatment Period 1: Adverse events occurring in the Placebo-Vasopressin group during the first 4-week treatment period (while receiving placebo).
- Placebo-Placebo Group - Treatment Period 1: Adverse events occurring in the Placebo-Placebo group during the first 4-week treatment period (while receiving placebo).
- Vasopressin-Vasopressin Group - Treatment Period 2: Adverse events occurring in the Vasopressin-Vasopressin group during the second 4-week treatment period (while receiving active drug).
- Placebo-Vasopressin Group - Treatment Period 2: Adverse events occurring in the Placebo-Vasopressin group during the second 4-week treatment period (while receiving active drug).
- Placebo-Placebo Group - Treatment Period 2: Adverse events occurring in the Placebo-Placebo group during the second 4-week treatment period (while receiving placebo).
- Open-label Vasopressin: Adverse events occurring in the Placebo-Placebo group during the open-label extension (after the 2 initial treatment periods, while receiving active drug).
Arm/Group | Vasopressin-Vasopressin Group - Treatment Period 1 | Placebo-Vasopressin Group - Treatment Period 1 | Placebo-Placebo Group - Treatment Period 1 | Vasopressin-Vasopressin Group - Treatment Period 2 | Placebo-Vasopressin Group - Treatment Period 2 | Placebo-Placebo Group - Treatment Period 2 | Open-label Vasopressin
Number analyzed (Participants) | 22 | 42 | 39 | 21 | 38 | 39 | 32
Participants
  Mild | 12 | 28 | 23 | 13 | 20 | 23 | 16
  Moderate | 3 | 15 | 18 | 5 | 13 | 13 | 9
  Severe | 0 | 1 | 0 | 1 | 0 | 2 | 1
  Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Death | 0 | 0 | 0 | 0 | 0 | 0 | 0

31. Other Pre Specified Outcome: Change From Baseline in Vineland Adaptive Behavior Scales, Third Edition (VABS-3) - Social Skills and Relationships Domain During Treatment.
Time Frame: 4-week; 8-week
Reporting Status: Not Posted

32. Other Pre Specified Outcome: Change From Baseline in Parent Rated Pediatric Quality of Life (PedsQL) Inventory Scores During Treatment.
Time Frame: 4-week; 8-week
Reporting Status: Not Posted

33. Other Pre Specified Outcome: Change From Baseline on Eye Gaze Assessment (Eye Tracking) During Treatment.
Time Frame: 4-week; 8-week
Reporting Status: Not Posted

34. Other Pre Specified Outcome: Change From Baseline on the Developmental Neuropsychological Assessment, Second Edition (NEPSY-II) Theory of Mind Test During Treatment.
Time Frame: 4-week; 8-week
Reporting Status: Not Posted

35. Other Pre Specified Outcome: Change From Baseline the Diagnostic Analysis of Nonverbal Accuracy, Second Edition (DANVA-2) Child Voices Prosody Test During Treatment.
Time Frame: 4-week; 8-week
Reporting Status: Not Posted

36. Other Pre Specified Outcome: Change From Baseline in Parent Rated Stanford Social Motivation Scale (Also Known as the Stanford Social Dimensional Scale) Total Scores During Treatment.
Time Frame: 4-week; 8-week
Reporting Status: Not Posted

37. Other Pre Specified Outcome: Change From Baseline in Parent Rated Anxiety Scale - Autism Spectrum Disorder (PRAS-ASD) Score During Treatment.
Time Frame: 4-week; 8-week
Reporting Status: Not Posted

38. Other Pre Specified Outcome: Change From Baseline in Parent Rated Social Responsiveness Scale, Second Edition (SRS-2) Social Avoidance Factor Score During Treatment.
Time Frame: 4-week; 8-week
Reporting Status: Not Posted

39. Other Pre Specified Outcome: Change From Baseline in Parent Rated Social Responsiveness Scale, Second Edition (SRS-2) Emotion Recognition Factor Score During Treatment.
Time Frame: 4-week; 8-week
Reporting Status: Not Posted

40. Other Pre Specified Outcome: Change From Baseline in Parent Rated Social Responsiveness Scale, Second Edition (SRS-2) Interpersonal Relatedness Factor Score During Treatment.
Time Frame: 4-week; 8-week
Reporting Status: Not Posted

41. Other Pre Specified Outcome: Change From Baseline in Parent Rated Social Responsiveness Scale, Second Edition (SRS-2) Insistence On Sameness Factor Score During Treatment.
Time Frame: 4-week; 8-week
Reporting Status: Not Posted

42. Other Pre Specified Outcome: Change From Baseline in Parent Rated Social Responsiveness Scale, Second Edition (SRS-2) Repetitive Mannerisms Factor Score During Treatment.
Time Frame: 4-week; 8-week
Reporting Status: Not Posted

43. Other Pre Specified Outcome: Change From Baseline in Parent Rated Social Responsiveness Scale, Second Edition (SRS-2) Attachment and Affiliation Factor Score During Treatment.
Time Frame: 4-week; 8-week
Reporting Status: Not Posted

44. Other Pre Specified Outcome: Change From Baseline in Parent Rated Social Responsiveness Scale, Second Edition (SRS-2) Non-facial Communication Production Factor Score During Treatment.
Time Frame: 4-week; 8-week
Reporting Status: Not Posted

45. Other Pre Specified Outcome: Change From Baseline in Parent Rated Social Responsiveness Scale, Second Edition (SRS-2) Facial Communication Production Factor Score During Treatment.
Time Frame: 4-week; 8-week
Reporting Status: Not Posted

46. Other Pre Specified Outcome: Change From Baseline in Parent Rated Social Responsiveness Scale, Second Edition (SRS-2) Mental States Understanding Factor Score During Treatment.
Time Frame: 4-week; 8-week
Reporting Status: Not Posted

47. Other Pre Specified Outcome: Change From Baseline in Parent Rated Child's Sleep Habits Questionnaire (CSHQ) Score During Treatment.
Time Frame: 4-week; 8-week
Reporting Status: Not Posted

48. Other Pre Specified Outcome: Change From Baseline on Spectral Power in the Alpha, Theta, and Gamma Frequencies as Measured by Electroencephalogram (EEG) During Treatment.
Time Frame: 4-week; 8-week
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: UP to 12 week
Arm/Group | Vasopressin-Vasopressin Group - Treatment Period 1 | Placebo-Vasopressin Group - Treatment Period 1 | Placebo-Placebo Group - Treatment Period 1 | Vasopressin-Vasopressin Group - Treatment Period 2 | Placebo-Vasopressin Group - Treatment Period 2 | Placebo-Placebo Group - Treatment Period 2 | Open-label Vasopressin
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/42 | 0/39 | 0/21 | 0/38 | 0/39 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/42 | 0/39 | 0/21 | 0/38 | 0/39 | 0/32
Other Adverse Events (participants affected / at risk) | 12/22 | 31/42 | 29/39 | 15/21 | 24/38 | 26/39 | 20/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vasopressin-Vasopressin Group - Treatment Period 1 (N=22) | Placebo-Vasopressin Group - Treatment Period 1 (N=42) | Placebo-Placebo Group - Treatment Period 1 (N=39) | Vasopressin-Vasopressin Group - Treatment Period 2 (N=21) | Placebo-Vasopressin Group - Treatment Period 2 (N=38) | Placebo-Placebo Group - Treatment Period 2 (N=39) | Open-label Vasopressin (N=32)
Dizziness (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1
Earache (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dilated Pupils (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye Redness (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eyelid Edema (Eye disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0
Hordeolum (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Lacrimation Increased (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 4 | 2 | 4 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 2 | 3 | 1 | 2 | 1 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0
Fecal Incontinence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flatuence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngeal Pain (Gastrointestinal disorders) | 1 | 2 | 5 | 2 | 0 | 0 | 2
Saliva Hypersecretion (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Throat Burning Sensation (Gastrointestinal disorders) | 0 | 3 | 1 | 0 | 1 | 1 | 0
Tooth Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting or Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 2 | 3 | 1
Pyrexia (General disorders) | 1 | 2 | 4 | 1 | 2 | 2 | 2
Seasonal Allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 3 | 1 | 1 | 2 | 0 | 0
Increased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Muscle Pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 0 | 0 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Agitation (Nervous system disorders) | 2 | 3 | 3 | 2 | 2 | 3 | 1
Headache (Nervous system disorders) | 2 | 4 | 3 | 0 | 5 | 4 | 4
Initial Insomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Middle Insomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Sedation (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 3 | 2 | 1 | 2 | 1 | 1
Unspecified Insomnia (Nervous system disorders) | 0 | 3 | 0 | 0 | 2 | 0 | 0
Aggression (Psychiatric disorders) | 1 | 8 | 10 | 5 | 8 | 7 | 8
Anal Picking (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Depressed Mood (Psychiatric disorders) | 1 | 1 | 2 | 2 | 1 | 1 | 1
Echopraxia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Finger Sucking (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperactivity (Psychiatric disorders) | 0 | 4 | 1 | 0 | 1 | 0 | 1
Impulsive Behavior (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Inappropriate Sexual Behavior (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Inattention (Psychiatric disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0
Irritability or Anger (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nail Biting (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Nightmares (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Psychomotor Retardation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Screaming (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Wandering Behavior (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Enuresis (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 5 | 1 | 2 | 6 | 1
Gag Reflex Abnormal (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 13 | 5 | 6 | 10 | 7
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1 | 1 | 1 | 1
Nasal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Nose Bleed (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3 | 1 | 0 | 2 | 0
Runny Nose (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4 | 2 | 2 | 0 | 0
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dysmenorrhea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Bug Bite (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 1 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 2 | 1 | 3 | 2 | 1
Scratch (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2020-03-27): https://cdn.clinicaltrials.gov/large-docs/86/NCT03204786/Prot_001.pdf
  • Statistical Analysis Plan (2023-11-17): https://cdn.clinicaltrials.gov/large-docs/86/NCT03204786/SAP_002.pdf
  • Informed Consent Form (2023-12-12): https://cdn.clinicaltrials.gov/large-docs/86/NCT03204786/ICF_000.pdf